CLINICAL TRIAL: NCT02890888
Title: The Effect of Hyperbaric Oxygen on the Functional Connectivity of Resting State Neural Networks in Patients With Cerebral Small Vessel Disease
Brief Title: Effect of Hyperbaric Oxygen on Functional Connectivity in Patients With Cerebral Small Vessel Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Depletion of Funds and Illness of principal investigator
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, John Davidson, Director, Division of Hyperbaric Medicine, St. Luke's Hospital, Chesterfield, Missouri
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.011
Record Dates: First submitted 2014-09-05; First posted 2016-09-07 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: small vessel disease of the brain; hyperbaric oxygen; functional connectivity MRI
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen treatment (Experimental): HBO for 1 hour at 2 ATA 10 times, administered 5 times per week over 2 consecutive weeks
  Interventions: Other: hyperbaric oxygen treatment

INTERVENTIONS:
Other: hyperbaric oxygen treatment — Patients are treated in a hyperbaric oxygen chamber for 1 hour at 2ATA, 10 times over 2 consecutive weeks, 5 times per week

SUMMARY:
Patients will have a Functional MRI before and after 10 hyperbaric Oxygen treatments.

DETAILED DESCRIPTION:
Functional MRI studies will be done before and 4-6 weeks after Hyperbaric Oxygen treatment to assess changes in connectivity of resting state neural networks. 10 hyperbaric treatments at 2 atmospheres absolute for 1 hour at pressure will be administered. A review of symptoms and and thorough clinical neurological examination by an experienced neurologist familiar with these studies will be done before and 4-6 weeks after the hyperbaric treatments.

ELIGIBILITY:
Inclusion Criteria:

* White Matter Hyperintensities on MRI
* 2 or more neurological symptoms or impairments e.g. gait disturbances, disequilibrium, cognitive decline, dysmetria, hyper-rflexia

Exclusion Criteria:

* Contraindication to hyperbaric oxygen treatment e.g. pulmonary emphysema, seizure disorder
* major eustachian tube dysfunction
* stroke with previous 6 months
* extreme cognitive impairment
* major depression
* history of migraine, electroshock therapy, brain irradiation, brain tumor, head trauma
* other uncontrolled co-morbidities, e.g. diabetes, renal or hepatic dysfunction, hypertension, thyroid disorders, carotid artery stenosis (>70%)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-11; Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Change in average functional connectivity (fc) within the Default Mode Network and the Dorsal Attention Network will be obtained by resting state network (rsn) functional connectivity (rsnfc) MRI. | Change in baseline rsnfc before and 4 weeks after hyperbaric oxygen
  Functional connectivity MRI of resting state neural networks.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Davidson, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - St. Luke's hospital, Chesterfield, Missouri
  - St. Luke's Hospital, St Louis, Missouri
  - Mallinckrodt Institute of Radiology/Washington University Medical School, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No